CLINICAL TRIAL: NCT02536339
Title: An Open-Label, Single-Arm, Phase II Study of Pertuzumab With High-Dose Trastuzumab for the Treatment of Central Nervous System Progression Post-Radiotherapy in Patients With HER2-Positive Metastatic Breast Cancer (PATRICIA)
Brief Title: A Study of Pertuzumab With High-Dose Trastuzumab for the Treatment of Human Epidermal Growth Factor Receptor 2 (HER2)-Positive Metastatic Breast Cancer (MBC) With Central Nervous System (CNS) Progression Post-Radiotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML29366
Record Dates: First submitted 2015-08-10; First posted 2015-08-31 (Estimated); Results first posted 2020-03-27 (Actual); Last update posted 2021-12-07 (Actual); Status verified 2021-12

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — pertuzumab; Trastuzumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pertuzumab + Trastuzumab (Experimental): Participants with CNS metastases secondary to HER2-positive MBC will receive pertuzumab in combination with high-dose trastuzumab until disease progression, unacceptable toxicity, withdrawal of consent, or study termination.
  Interventions: Drug: Pertuzumab; Drug: Trastuzumab

INTERVENTIONS:
Drug: Pertuzumab — Participants will receive 840 milligrams (mg) loading dose of pertuzumab, followed every 3 weeks thereafter by a dose of 420 mg via intravenous (IV) infusion until disease progression, unacceptable toxicity, withdrawal of consent, or study termination.
  Other Names: Perjeta; RO4368451
Drug: Trastuzumab — Participants will receive trastuzumab at a dose of 6 milligrams per kilogram (mg/kg) of body weight once weekly via IV infusion until disease progression, unacceptable toxicity, withdrawal of consent, or study termination.
  Other Names: Herceptin; RO0452317

SUMMARY:
This study will examine the safety and efficacy of pertuzumab in combination with high-dose trastuzumab in adult participants with HER2-positive MBC with CNS metastases and disease progression in the brain following radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed HER2-positive MBC
* Progression of or new brain metastases after completion of whole-brain radiotherapy or stereotactic radiosurgery
* Completion of whole-brain radiotherapy or stereotactic radiosurgery more than 60 days prior to enrollment
* Stable systemic disease
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* LVEF at least 50%
* Adequate hematologic, renal, and hepatic function
* Life expectancy more than 12 weeks

Exclusion Criteria:

* Progression of systemic disease at Screening
* Leptomeningeal disease
* History of intolerance or hypersensitivity to study drug
* Use of certain investigational therapies within 21 days prior to enrollment
* Current anthracycline use
* Unwillingness to discontinue ado-trastuzumab emtansine or lapatinib use
* Active infection
* Pregnant or lactating women
* Significant history or risk of cardiac disease
* Symptomatic intrinsic lung disease or lung involvement
* History of other malignancy within the last 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-12-16 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2020-12-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (16):
- United States (16):
  - Arizona Cancer Center, Tucson, Arizona
  - City of Hope National Medical Center, Duarte, California
  - Stanford Cancer Institute, Stanford, California
  - University of Miami Hospital & Clinics, Miami, Florida
  - H. Lee Moffitt Cancer Center and Research Inst., Tampa, Florida
  - Northwestern University, Chicago, Illinois
  - University of Maryland Medical Center; Department of Neurology, Baltimore, Maryland
  - Associates in Oncology-Hematology, PC, Bethesda, Maryland
  - Dana Farber Cancer Inst., Boston, Massachusetts
  - Allina Health System, Saint Paul, Minnesota
  - Stony Brook University Medical Center, Stony Brook, New York
  - Mid Ohio Oncology Hematology;ZangMeister Center (West), Columbus, Ohio
  - Temple Cancer Center; Oncology, Philadelphia, Pennsylvania
  - Methodist Hospital Research Institute, Houston, Texas
  - Huntsman Cancer Institute; University of Utah, Salt Lake City, Utah
  - Northwest Medical Specialties, PLLC, Tacoma, Washington

REFERENCES:
- [Derived] Lin NU, Pegram M, Sahebjam S, Ibrahim N, Fung A, Cheng A, Nicholas A, Kirschbrown W, Kumthekar P. Pertuzumab Plus High-Dose Trastuzumab in Patients With Progressive Brain Metastases and HER2-Positive Metastatic Breast Cancer: Primary Analysis of a Phase II Study. J Clin Oncol. 2021 Aug 20;39(24):2667-2675. doi: 10.1200/JCO.20.02822. Epub 2021 May 4. PMID 33945296

RESULTS

PARTICIPANT FLOW:
Groups:
- Pertuzumab + Trastuzumab: Participants with CNS metastases secondary to HER2-positive MBC, who had disease progression in the brain following previous treatment with radiotherapy (whole-brain radiation therapy or stereotactic radiosurgery) for brain metastases, received treatment with pertuzumab in combination with high-dose trastuzumab until disease progression, unacceptable toxicity, withdrawal of consent, or study termination by the Sponsor, whichever occurred first.
Period: Overall Study
Arm/Group | Pertuzumab + Trastuzumab
Started (Intention-to-Treat (ITT) Population) | 40
Received at Least One Dose of Study Drug (Safety Population) | 39
Efficacy-Evaluable Population | 37 (2 participants did not have post-baseline assessments and were not evaluable for efficacy.)
Completed | 12
Not Completed | 28
Not completed — Death | 20
Not completed — Withdrawal by Subject | 3
Not completed — Lost to Follow-up | 2
Not completed — Treatment discontinued | 2
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) population: all enrolled patients in the study, regardless of whether they were exposed to study treatment.
Arm/Group | Pertuzumab + Trastuzumab
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50.0 (9.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 33
  Unknown or Not Reported | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 36
  Asian | 2
  Other Race | 1
  Not Reported | 1
Women of Childbearing Potential Status [Count of Participants; unit: Participants]
  Childbearing Potential | 12
  Non-Childbearing Potential - Postmenopausal | 21
  Non-Childbearing Potential - Surgically Sterile | 7
Left Ventricular Ejection Fraction (LVEF) Value at Baseline [Median (Full Range); unit: Percentage Points of LVEF (%)] — Population: The LVEF analysis was performed on the safety analysis population, which included all participants who received at least one dose of study treatment. One participant who did not receive any study drug was excluded from the analysis.
  Percentage Points of LVEF (%)
    number analyzed (Participants) | 39
    (all) | 60.00 [50.00 to 75.00]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Objective Response in the CNS, Assessed Using Response Assessment in Neuro-Oncology-Brain Metastases (RANO-BM) Criteria
Description: Responses were assessed by the investigator, based on magnetic resonance imaging (MRI) of the brain, physical examinations, routine neurological examinations, and corticosteroid dosing. An objective response in the central nervous system (CNS) was a complete response (CR) or partial response (PR) confirmed by repeat assessment, according to RANO-BM criteria. A CR was defined as the disappearance of all CNS target lesions sustained for at least 4 weeks; no new lesions; no corticosteroids; and stable or improved clinically; for non-target lesions, a CR was the disappearance of all enhancing CNS non-target lesions and no new CNS lesions. A PR was defined as at least a 30% decrease in the sum longest diameter (LD) of CNS target lesions, taking as reference the baseline sum LD sustained for at least 4 weeks; no new lesions; stable to decreased corticosteroid dose; and stable or improved clinically. The 95% Clopper-Pearson exact confidence intervals were calculated for responses.
Time Frame: From Baseline until disease progression (assessed every 6 weeks for first 2 scans, followed by every 8 weeks for 2 scans, then every 12 weeks until disease progression; up to approximately 3.5 years)
Population: Efficacy-Evaluable Population: all participants who received any dose of study treatment and had at least one follow-up CNS tumor assessment or died without follow-up tumor assessment within 30 days from the last dose of study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pertuzumab + Trastuzumab
Number analyzed (Participants) | 37
Percentage of Participants
  With Objective Response (Confirmed CR or PR) | 10.8 [3.03 to 25.42]
  Confirmed Complete Response (CR) | 0.0 [0.00 to 9.49]
  Confirmed Partial Response (PR) | 10.8 [3.03 to 25.42]
  Without Objective Response | 89.2 [NA to NA] — The 95% confidence intervals were only calculated for objective responses.

2. Secondary Outcome: Median Duration of Response in the CNS, Assessed Using RANO-BM Criteria
Description: Responses were assessed by the investigator, based on magnetic resonance imaging (MRI) of the brain, physical examinations, routine neurological examinations, and corticosteroid dosing. An objective response in the central nervous system (CNS) was a complete response (CR) or partial response (PR) confirmed by repeat assessment, according to RANO-BM criteria. Among participants who achieved an objective response, duration of response in the CNS was defined as the time from documentation of the first CR or PR to the time of disease progression, relapse, or death from any cause. If a participant did not experience death or disease progression in the CNS before the end of the study, duration of response was censored on the last date the participant was known to be progression free. Duration of response was estimated by the Kaplan-Meier method.
Time Frame: From documentation of first complete response (CR) or partial response (PR) to the time of disease progression, relapse, or death from any cause, whichever occurred first (up to approximately 3.5 years)
Population: Efficacy-Evaluable Population: all participants who received any dose of study treatment and had at least one follow-up CNS tumor assessment or died without follow-up tumor assessment within 30 days from the last dose of study treatment. Only participants who had a confirmed CR or PR in the CNS were included in this analysis.
Measure: Median (Full Range); unit: Months
Arm/Group | Pertuzumab + Trastuzumab
Number analyzed (Participants) | 4
Months | 4.60 [3.19 to 5.59]

3. Secondary Outcome: Percentage of Participants With Clinical Benefit (Confirmed CR, PR, or Stable Disease [SD] ≥4 Months) in the CNS, Assessed Using RANO-BM Criteria
Description: Responses were assessed by the investigator, based on magnetic resonance imaging (MRI) of the brain, physical examinations, routine neurological examinations, and corticosteroid dosing. Clinical benefit in the central nervous system (CNS) was defined here as a complete response (CR), partial response (PR), or stable disease (SD) for at least 4 months, confirmed by repeat assessment according to RANO-BM criteria. A CR or PR were defined in the same way as for objective response in the CNS. SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum longest diameter (LD) while on study. The 95% Clopper-Pearson exact confidence intervals were calculated for responses.
Time Frame: From Baseline until disease progression (assessed every 6 weeks for first 2 scans, followed by every 8 weeks for 2 scans, then every 12 weeks until disease progression; up to approximately 5 years)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pertuzumab + Trastuzumab
Number analyzed (Participants) | 37
Percentage of Participants
  With Clinical Benefit (Confirmed CR,PR,or SD≥4mos) | 67.6 [50.21 to 81.99]
  Confirmed Complete Response (CR) | 0.0 [0.00 to 9.49]
  Confirmed Partial Response (PR) | 10.8 [3.03 to 25.42]
  Confirmed Stable Disease (SD) ≥4 Months | 56.8 [39.49 to 72.90]
  Without Clinical Benefit | 32.4 [NA to NA] — The 95% confidence intervals were only calculated for clinical benefit responses.

4. Secondary Outcome: Median Duration of Clinical Benefit (Confirmed CR, PR, or SD ≥4 Months) in the CNS, Assessed Using RANO-BM Criteria
Description: Responses were assessed by the investigator, based on magnetic resonance imaging (MRI) of the brain, physical examinations, routine neurological examinations, and corticosteroid dosing. Clinical benefit in the central nervous system (CNS) was defined here as a complete response (CR), partial response (PR), or stable disease (SD) for at least 4 months, confirmed by repeat assessment according to RANO-BM criteria. Among participants who achieved clinical benefit, duration of clinical benefit in the CNS was defined as the time from documentation of the first CR, PR, or SD ≥4 months to the time of disease progression, relapse, or death from any cause. If a participant did not experience death or disease progression in the CNS before the end of the study, duration of clinical benefit was censored on the last date the participant was known to be progression free. Duration of clinical benefit was estimated by the Kaplan-Meier method.
Time Frame: From documentation of first complete response (CR), partial response (PR), or stable disease (SD) ≥4 months to the date of disease progression, relapse, or death from any cause, whichever occurred first (up to approximately 5 years)
Population: Efficacy-Evaluable Population: all participants who received any dose of study treatment and had at least one follow-up CNS tumor assessment or died without follow-up tumor assessment within 30 days from the last dose of study treatment. Only those with confirmed CR, PR, or SD ≥4 months in the CNS were included in this analysis.
Measure: Median (Full Range); unit: Months
Arm/Group | Pertuzumab + Trastuzumab
Number analyzed (Participants) | 25
Months | 6.64 [3.2 to 56.1]

5. Secondary Outcome: Percentage of Participants With Clinical Benefit (Confirmed CR, PR, or SD ≥6 Months) in the CNS, Assessed Using RANO-BM Criteria
Description: Responses were assessed by the investigator, based on magnetic resonance imaging (MRI) of the brain, physical examinations, routine neurological examinations, and corticosteroid dosing. Clinical benefit in the central nervous system (CNS) was defined here as a complete response (CR), partial response (PR), or stable disease (SD) for at least 6 months, confirmed by repeat assessment according to RANO-BM criteria. A CR or PR were defined in the same way as for objective response in the CNS. SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum longest diameter (LD) while on study. The 95% Clopper-Pearson exact confidence intervals were calculated for responses.
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pertuzumab + Trastuzumab
Number analyzed (Participants) | 37
Percentage of Participants
  With Clinical Benefit (Confirmed CR,PR,or SD≥6mos) | 51.4 [34.40 to 68.08]
  Confirmed Complete Response (CR) | 0.0 [0.00 to 9.49]
  Confirmed Partial Response (PR) | 10.8 [3.03 to 25.42]
  Confirmed Stable Disease (SD) ≥6 Months | 40.5 [24.75 to 57.90]
  Without Clinical Benefit | 48.6 [NA to NA] — The 95% confidence intervals were only calculated for clinical benefit responses.

6. Secondary Outcome: Median Duration of Clinical Benefit (Confirmed CR, PR, or SD ≥6 Months) in the CNS, Assessed Using RANO-BM Criteria
Description: Responses were assessed by the investigator, based on magnetic resonance imaging (MRI) of the brain, physical examinations, routine neurological examinations, and corticosteroid dosing. Clinical benefit in the central nervous system (CNS) was defined here as a complete response (CR), partial response (PR), or stable disease (SD) for at least 6 months, confirmed by repeat assessment according to RANO-BM criteria. Among participants who achieved clinical benefit, duration of clinical benefit in the CNS was defined as the time from documentation of the first CR, PR, or SD ≥6 months to the time of disease progression, relapse, or death from any cause. If a participant did not experience death or disease progression in the CNS before the end of the study, duration of clinical benefit was censored on the last date the participant was known to be progression free. Duration of clinical benefit was estimated by the Kaplan-Meier method.
Time Frame: From documentation of first complete response (CR), partial response (PR), or stable disease (SD) ≥6 months to the date of disease progression, relapse, or death from any cause, whichever occurred first (up to approximately 5 years)
Population: Efficacy-Evaluable Population: all participants who received any dose of study treatment and had at least one follow-up CNS tumor assessment or died without follow-up tumor assessment within 30 days from the last dose of study treatment. Only those with confirmed CR, PR, or SD ≥6 months in the CNS were included in this analysis.
Measure: Median (Full Range); unit: Months
Arm/Group | Pertuzumab + Trastuzumab
Number analyzed (Participants) | 19
Months | 9.23 [3.2 to 56.1]

7. Secondary Outcome: Progression-Free Survival (CNS), Assessed Using RANO-BM Criteria
Description: Progression-free survival (CNS) was defined as the time from the date of first dose to disease progression in the CNS or death from any cause. If no progressive disease in the CNS and no death occurred, progression-free survival (CNS) was censored on the date of the last CNS tumor assessment. If a post-baseline assessment was not available, progression-free survival (CNS) was censored on Day 1.
Time Frame: From the date of first dose to disease progression in the CNS or death from any cause, whichever occurred first (up to approximately 5 years)
Population: as for outcome 1
Measure: Median (Full Range); unit: Months
Arm/Group | Pertuzumab + Trastuzumab
Number analyzed (Participants) | 37
Months | 4.63 [0.82 to 56.11]

8. Secondary Outcome: Progression-Free Survival (Systemic), Assessed Using Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST v1.1)
Description: Progression-free survival (systemic) was defined as the time from the date of first dose to systemic disease progression or death from any cause. If no systemic disease progression and no death occurred, progression-free survival (systemic) was censored on the date of the last systemic tumor assessment. If a post-baseline assessment was not available, progression-free survival (systemic) was censored on Day 1.
Time Frame: From the date of first dose to systemic disease progression or death from any cause, whichever occurred first (up to approximately 5 years)
Population: as for outcome 1
Measure: Median (Full Range); unit: Months
Arm/Group | Pertuzumab + Trastuzumab
Number analyzed (Participants) | 37
Months | 16.26 [0.03 to 55.20]

9. Secondary Outcome: Progression-Free Survival (CNS or Systemic), Assessed Using RANO-BM Criteria and RECIST v1.1
Description: Progression-free survival (CNS or systemic) was defined as the time from the date of first dose to CNS or systemic disease progression or death from any cause. If no CNS or systemic disease progression and no death occurred, data was censored on the date of the last CNS or systemic tumor assessment, whichever occurred first. If a post-baseline assessment was not available, data was censored on Day 1.
Time Frame: From the date of first dose to CNS or systemic disease progression or death from any cause, whichever occurred first (up to approximately 5 years)
Population: as for outcome 1
Measure: Median (Full Range); unit: Months
Arm/Group | Pertuzumab + Trastuzumab
Number analyzed (Participants) | 37
Months | 4.63 [0.03 to 55.20]

10. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the period from the date of first dose until the date of death from any cause. If no death occurred, overall survival was censored on the last date the participant was known to be alive.
Time Frame: From the date of first dose until death due to any cause (up to approximately 5 years)
Population: as for outcome 1
Measure: Median (Full Range); unit: Months
Arm/Group | Pertuzumab + Trastuzumab
Number analyzed (Participants) | 37
Months | 27.17 [0.82 to 57.49]

11. Secondary Outcome: Number of Deaths by Time (≤30 or >30 Days) From Last Study Drug Administration and by Primary Cause of Death
Time Frame: From date of first dose until death due to any cause (up to approximately 5 years)
Population: Safety Population: all participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pertuzumab + Trastuzumab
Number analyzed (Participants) | 39
Participants
  All Deaths | 20
  Deaths ≤30 Days From Last Dose of Study Drug | 1
  Deaths >30 Days From Last Dose of Study Drug | 19
  Primary Cause of Death: Progressive Disease | 16
  Primary Cause of Death: Other Cause (and Cancer) | 1
  Primary Cause of Death: Unknown | 3

12. Secondary Outcome: Number of Participants With at Least One Treatment-Emergent Adverse Event (TEAE) by Highest Grade of Severity, According to National Cancer Institute Common Terminology Criteria for Adverse Events, Version 4.0 (NCI-CTCAE v4.0)
Description: Treatment-emergent adverse events (TEAEs) were defined as all adverse events occurring on or after Day 1 of study treatment until 30 days after the last dose of study treatment. All TEAEs were graded for severity using the NCI-CTCAE v4.0; any TEAE not specifically listed was assessed per the following 5 grades: Grade 1 = mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; or intervention not indicated. Grade 2 = moderate; minimal, local, or non-invasive intervention indicated; or limiting age-appropriate instrumental activities of daily living. Grade 3 = severe or medically significant, but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; or limiting self-care activities of daily living. Grade 4 = life-threatening consequences or urgent intervention indicated. Grade 5 = death related to adverse event. Multiple occurrences of TEAEs were counted only once per participant at the highest (worst) grade.
Time Frame: From the first dose until 30 days after the last dose of study treatment (up to approximately 5 years)
Population: Safety Population: all participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pertuzumab + Trastuzumab
Number analyzed (Participants) | 39
Participants
  Any TEAE - Any Grade | 38
  Any TEAE - Grade 1 | 5
  Any TEAE - Grade 2 | 16
  Any TEAE - Grade 3 | 14
  Any TEAE - Grade 4 | 3
  Any TEAE - Grade 5 | 0

13. Secondary Outcome: Number of Participants With at Least One Treatment-Emergent Serious Adverse Event (SAE) by Highest Grade of Severity, According to NCI-CTCAE v4.0
Description: Treatment-emergent serious adverse events (SAEs) were defined as all adverse events that met seriousness criteria (as defined in the protocol; same as the ClinicalTrials.gov definition) occurring on or after Day 1 of study treatment until 30 days after the last dose of study treatment. All SAEs were graded for severity using the NCI-CTCAE v4.0; any SAE not specifically listed was assessed per the following 5 grades: Grade 1 = mild; Grade 2 = moderate; Grade 3 = severe or medically significant, but not immediately life-threatening; Grade 4 = life-threatening consequences or urgent intervention indicated; and Grade 5 = death related to adverse event. The terms "severe" and "serious" are not synonymous and are independently assessed for each adverse event. Multiple occurrences of SAEs were counted only once per participant at the highest (worst) grade.
Time Frame: From the first dose until 30 days after the last dose of study treatment (up to approximately 5 years)
Population: Safety Population: all participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pertuzumab + Trastuzumab
Number analyzed (Participants) | 39
Participants
  Any SAE - Any Grade | 7
  Any SAE - Grade 1 | 0
  Any SAE - Grade 2 | 1
  Any SAE - Grade 3 | 5
  Any SAE - Grade 4 | 2
  Any SAE - Grade 5 | 0

14. Secondary Outcome: Number of Participants With at Least One TEAE Leading to Withdrawal of Any Study Drug, Pertuzumab Only, or Both Pertuzumab and Trastuzumab, by Highest Grade of Severity According to NCI-CTCAE v4.0
Description: as for outcome 12
Time Frame: From the first dose until 30 days after the last dose of study treatment (up to approximately 5 years)
Population: Safety Population: all participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pertuzumab + Trastuzumab
Number analyzed (Participants) | 39
Participants
  Withdrawal of Any Study Drug - Any Grade TEAE | 2
  Withdrawal of Any Study Drug - Grade 3 TEAE | 2
  Withdrawal of Pertuzumab Only - Any Grade TEAE | 0
  Withdrawal of Both Study Drugs - Any Grade TEAE | 2
  Withdrawal of Both Study Drugs - Grade 3 TEAE | 2

15. Secondary Outcome: Number of Participants With at Least One TEAE Leading to Pertuzumab Infusion Delay, Slow Down, or Interruption, by Highest Grade of Severity According to NCI-CTCAE v4.0
Description: as for outcome 12
Time Frame: From the first dose until 30 days after the last dose of study treatment (up to approximately 5 years)
Population: Safety Population: all participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pertuzumab + Trastuzumab
Number analyzed (Participants) | 39
Participants
  Any TEAE - Any Grade | 7
  Any TEAE - Grade 1 | 1
  Any TEAE - Grade 2 | 4
  Any TEAE - Grade 3 | 1
  Any TEAE - Grade 4 | 1
  Any TEAE - Grade 5 | 0

16. Secondary Outcome: Number of Participants With at Least One TEAE Leading to Trastuzumab Dose Modification by Highest Grade of Severity According to NCI-CTCAE v4.0
Description: as for outcome 12
Time Frame: From the first dose until 30 days after the last dose of study treatment (up to approximately 5 years)
Population: Safety Population: all participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pertuzumab + Trastuzumab
Number analyzed (Participants) | 39
Participants
  Any TEAE - Any Grade | 12
  Any TEAE - Grade 1 | 2
  Any TEAE - Grade 2 | 4
  Any TEAE - Grade 3 | 5
  Any TEAE - Grade 4 | 1
  Any TEAE - Grade 5 | 0

17. Secondary Outcome: Percentage of Participants With at Least One TEAE of Special Interest by Highest Grade of Severity, According to NCI-CTCAE v4.0
Description: Protocol-defined TEAEs of special interest, occurring on or after Day 1 of study treatment until 30 days after the last dose of study treatment, included the following: An elevated ALT or AST (>3 times baseline value) in combination with either an elevated total bilirubin (>2 times the upper limit of normal) or clinical jaundice; Suspected transmission of an infectious agent by the study treatment; Congestive heart failure; An asymptomatic decline in LVEF (a value 10 percentage points below baseline or lower, and <45%) that requires treatment or that leads to discontinuation of study treatment. All TEAEs of special interest were graded for severity using the NCI-CTCAE v4.0. Multiple occurrences of TEAEs of special interest were counted only once per participant at the highest (worst) grade.
Time Frame: From the first dose until 30 days after the last dose of study treatment (up to approximately 5 years)
Population: Safety Population: all participants who received at least one dose of study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pertuzumab + Trastuzumab
Number analyzed (Participants) | 39
Percentage of Participants
  Any TEAE of Special Interest - Any Grade | 2.6 [0.06 to 13.48]
  Asymptomatic Decline in LVEF - Grade 3 | 2.6 [0.06 to 13.48]

18. Secondary Outcome: Median Left Ventricular Ejection Fraction (LVEF) Values Over Time
Description: Left ventricular ejection fraction (LVEF) is the measurement of the percentage of blood that is being pumped out of the left ventricle of the heart (the main pumping chamber) with each contraction. All participants were required to have had a baseline LVEF of at least 50% to participate in this study. Measurements were done by either echocardiogram (ECHO) or mulitple-gated acquisition (MUGA) scan (with ECHO as the preferred method). Participants were to be reassessed with the same technique used for baseline cardiac evaluation throughout the study.
Time Frame: Baseline, Weeks 6, 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, and 132 (Treatment Period); and every 3 months during Survival Follow-Up (up to approximately 5 years)
Population: Safety Population: all participants who received at least one dose of study treatment. Only participants with evaluable assessments at each visit were included in the analysis.
Measure: Median (Full Range); unit: Percentage Points of LVEF (%)
Arm/Group | Pertuzumab + Trastuzumab
Number analyzed (Participants) | 39
Percentage Points of LVEF (%)
  Baseline | 60.00 [50.00 to 75.00]
  Week 6: number analyzed (Participants) | 34
  Week 6 | 60.00 [30.00 to 69.00]
  Week 12: number analyzed (Participants) | 30
  Week 12 | 60.00 [51.00 to 73.00]
  Week 24: number analyzed (Participants) | 15
  Week 24 | 60.00 [50.00 to 67.00]
  Week 36: number analyzed (Participants) | 9
  Week 36 | 60.00 [50.00 to 65.00]
  Week 48: number analyzed (Participants) | 7
  Week 48 | 60.00 [48.00 to 64.00]
  Week 60: number analyzed (Participants) | 7
  Week 60 | 62.00 [49.00 to 70.00]
  Week 72: number analyzed (Participants) | 4
  Week 72 | 55.50 [53.00 to 65.00]
  Week 84: number analyzed (Participants) | 3
  Week 84 | 60.00 [55.00 to 62.00]
  Week 96: number analyzed (Participants) | 3
  Week 96 | 63.00 [60.00 to 65.00]
  Week 108: number analyzed (Participants) | 2
  Week 108 | 62.00 [60.00 to 64.00]
  Week 120: number analyzed (Participants) | 1
  Week 120 | 64.00 [64.00 to 64.00]
  Week 132: number analyzed (Participants) | 1
  Week 132 | 64.00 [64.00 to 64.00]
  Survival Follow-Up 1: number analyzed (Participants) | 5
  Survival Follow-Up 1 | 60.00 [50.00 to 68.00]
  Survival Follow-Up 2: number analyzed (Participants) | 12
  Survival Follow-Up 2 | 59.00 [53.00 to 75.00]
  Survival Follow-Up 3: number analyzed (Participants) | 5
  Survival Follow-Up 3 | 60.00 [55.00 to 65.00]
  Survival Follow-Up 4: number analyzed (Participants) | 2
  Survival Follow-Up 4 | 69.00 [66.00 to 72.00]
  Survival Follow-Up 5: number analyzed (Participants) | 3
  Survival Follow-Up 5 | 67.00 [60.00 to 72.00]
  Survival Follow-Up 6: number analyzed (Participants) | 3
  Survival Follow-Up 6 | 57.00 [55.00 to 58.00]
  Survival Follow-Up 7: number analyzed (Participants) | 2
  Survival Follow-Up 7 | 57.50 [55.00 to 60.00]
  Survival Follow-Up 8: number analyzed (Participants) | 2
  Survival Follow-Up 8 | 57.00 [55.00 to 59.00]

19. Secondary Outcome: Number of Participants by Investigator Interpretation of Left Ventricular Ejection Fraction (LVEF) Assessments Over Time
Description: Left ventricular ejection fraction (LVEF) is the measurement of the percentage of blood that is being pumped out of the left ventricle of the heart (the main pumping chamber) with each contraction. All participants were required to have had a baseline LVEF of at least (≥)50% to participate in this study. Measurements were done by either echocardiogram (ECHO) or mulitple-gated acquisition (MUGA) scan (with ECHO as the preferred method). Participants were to be reassessed with the same technique used for baseline cardiac evaluation throughout the study. The following are definitions for the three categories of LVEF findings: 'Normal' was defined as LVEF >45% or LVEF 40-45% with less than (<)10% points drop below baseline; 'Abnormal' was defined as LVEF <40% or LVEF ≥10% points drop below baseline, and clinically significant versus non-clinically significant was subject to the investigator's assessment of whether symptoms were present or absent.
Time Frame: as for outcome 18
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | Pertuzumab + Trastuzumab
Number analyzed (Participants) | 39
Participants
  Baseline: Normal | 39
  Baseline: Abnormal, Not Clinically Significant | 0
  Baseline: Abnormal, Clinically Significant | 0
  Week 6: number analyzed (Participants) | 34
  Week 6: Normal | 33
  Week 6: Abnormal, Not Clinically Significant | 0
  Week 6: Abnormal, Clinically Significant | 1
  Week 12: number analyzed (Participants) | 30
  Week 12: Normal | 30
  Week 12: Abnormal, Not Clinically Significant | 0
  Week 12: Abnormal, Clinically Significant | 0
  Week 24: number analyzed (Participants) | 15
  Week 24: Normal | 14
  Week 24: Abnormal, Not Clinically Significant | 1
  Week 24: Abnormal, Clinically Significant | 0
  Week 36: number analyzed (Participants) | 9
  Week 36: Normal | 9
  Week 36: Abnormal, Not Clinically Significant | 0
  Week 36: Abnormal, Clinically Significant | 0
  Week 48: number analyzed (Participants) | 7
  Week 48: Normal | 6
  Week 48: Abnormal, Not Clinically Significant | 1
  Week 48: Abnormal, Clinically Significant | 0
  Week 60: number analyzed (Participants) | 7
  Week 60: Normal | 6
  Week 60: Abnormal, Not Clinically Significant | 1
  Week 60: Abnormal, Clinically Significant | 0
  Week 72: number analyzed (Participants) | 4
  Week 72: Normal | 4
  Week 72: Abnormal, Not Clinically Significant | 0
  Week 72: Abnormal, Clinically Significant | 0
  Week 84: number analyzed (Participants) | 3
  Week 84: Normal | 3
  Week 84: Abnormal, Not Clinically Significant | 0
  Week 84: Abnormal, Clinically Significant | 0
  Week 96: number analyzed (Participants) | 3
  Week 96: Normal | 3
  Week 96: Abnormal, Not Clinically Significant | 0
  Week 96: Abnormal, Clinically Significant | 0
  Week 108: number analyzed (Participants) | 2
  Week 108: Normal | 2
  Week 108: Abnormal, Not Clinically Significant | 0
  Week 108: Abnormal, Clinically Significant | 0
  Week 120: number analyzed (Participants) | 1
  Week 120: Normal | 1
  Week 120: Abnormal, Not Clinically Significant | 0
  Week 120: Abnormal, Clinically Significant | 0
  Week 132: number analyzed (Participants) | 1
  Week 132: Normal | 1
  Week 132: Abnormal, Not Clinically Significant | 0
  Week 132: Abnormal, Clinically Significant | 0
  Survival Follow-Up 1: number analyzed (Participants) | 5
  Survival Follow-Up 1: Normal | 5
  Survival Follow-Up 1: Abnormal, Not Clinically Significant | 0
  Survival Follow-Up 1: Abnormal, Clinically Significant | 0
  Survival Follow-Up 2: number analyzed (Participants) | 12
  Survival Follow-Up 2: Normal | 12
  Survival Follow-Up 2: Abnormal, Not Clinically Significant | 0
  Survival Follow-Up 2: Abnormal, Clinically Significant | 0
  Survival Follow-Up 3: number analyzed (Participants) | 5
  Survival Follow-Up 3: Normal | 5
  Survival Follow-Up 3: Abnormal, Not Clinically Significant | 0
  Survival Follow-Up 3: Abnormal, Clinically Significant | 0
  Survival Follow-Up 4: number analyzed (Participants) | 2
  Survival Follow-Up 4: Normal | 1
  Survival Follow-Up 4: Abnormal, Not Clinically Significant | 1
  Survival Follow-Up 4: Abnormal, Clinically Significant | 0
  Survival Follow-Up 5: number analyzed (Participants) | 3
  Survival Follow-Up 5: Normal | 3
  Survival Follow-Up 5: Abnormal, Not Clinically Significant | 0
  Survival Follow-Up 5: Abnormal, Clinically Significant | 0
  Survival Follow-Up 6: number analyzed (Participants) | 3
  Survival Follow-Up 6: Normal | 3
  Survival Follow-Up 6: Abnormal, Not Clinically Significant | 0
  Survival Follow-Up 6: Abnormal, Clinically Significant | 0
  Survival Follow-Up 7: number analyzed (Participants) | 2
  Survival Follow-Up 7: Normal | 2
  Survival Follow-Up 7: Abnormal, Not Clinically Significant | 0
  Survival Follow-Up 7: Abnormal, Clinically Significant | 0
  Survival Follow-Up 8: number analyzed (Participants) | 2
  Survival Follow-Up 8: Normal | 2
  Survival Follow-Up 8: Abnormal, Not Clinically Significant | 0
  Survival Follow-Up 8: Abnormal, Clinically Significant | 0

20. Secondary Outcome: Number of Participants With NCI-CTCAE v4.0 Grades 3 and 4 Clinical Laboratory Abnormalities in Hematology Tests Over Time
Description: Clinical laboratory tests for hematology parameters were performed every 6 weeks and any abnormal values (High or Low) were based on NCI-CTCAE v4.0 grades. Laboratory abnormalities of NCI-CTCAE v4.0 Grades 3 and 4 are presented. Not every abnormal laboratory value qualified as an adverse event, only if it met any of the following criteria: clinically significant (per investigator); accompanied by clinical symptoms; resulted in a change in study treatment; or required a change in concomitant therapy. For the overall category, multiple occurrences of the same laboratory abnormality over time in one participant were only counted once.
Time Frame: Baseline, Weeks 18, 36, and 60 (up to approximately 5 years)
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | Pertuzumab + Trastuzumab
Number analyzed (Participants) | 39
Participants
  Overall: Lymphocytes (10^9/L), Low - Grade 3: number analyzed (Participants) | 36
  Overall: Lymphocytes (10^9/L), Low - Grade 3 | 3
  Overall: Lymphocytes (10^9/L), High - Grade 3: number analyzed (Participants) | 36
  Overall: Lymphocytes (10^9/L), High - Grade 3 | 0
  Overall: Lymphocytes (10^9/L), Low - Grade 4: number analyzed (Participants) | 36
  Overall: Lymphocytes (10^9/L), Low - Grade 4 | 1
  Overall: Lymphocytes (10^9/L), High - Grade 4: number analyzed (Participants) | 36
  Overall: Lymphocytes (10^9/L), High - Grade 4 | 0
  Baseline: Lymphocytes (10^9/L), Low - Grade 3: number analyzed (Participants) | 35
  Baseline: Lymphocytes (10^9/L), Low - Grade 3 | 2
  Baseline: Lymphocytes (10^9/L), Low - Grade 4: number analyzed (Participants) | 35
  Baseline: Lymphocytes (10^9/L), Low - Grade 4 | 0
  Week 18: Lymphocytes (10^9/L), Low - Grade 3: number analyzed (Participants) | 20
  Week 18: Lymphocytes (10^9/L), Low - Grade 3 | 1
  Week 18: Lymphocytes (10^9/L), Low - Grade 4: number analyzed (Participants) | 20
  Week 18: Lymphocytes (10^9/L), Low - Grade 4 | 0
  Week 36: Lymphocytes (10^9/L), Low - Grade 3: number analyzed (Participants) | 8
  Week 36: Lymphocytes (10^9/L), Low - Grade 3 | 1
  Week 36: Lymphocytes (10^9/L), Low - Grade 4: number analyzed (Participants) | 8
  Week 36: Lymphocytes (10^9/L), Low - Grade 4 | 0
  Week 60: Lymphocytes (10^9/L), Low - Grade 3: number analyzed (Participants) | 7
  Week 60: Lymphocytes (10^9/L), Low - Grade 3 | 0
  Week 60: Lymphocytes (10^9/L), Low - Grade 4: number analyzed (Participants) | 7
  Week 60: Lymphocytes (10^9/L), Low - Grade 4 | 1

21. Secondary Outcome: Number of Participants With NCI-CTCAE v4.0 Grades 3 and 4 Clinical Laboratory Abnormalities in Blood Chemistry Tests Over Time
Description: Clinical laboratory tests for blood chemistry parameters were performed every 6 weeks and any abnormal values (High or Low) were based on NCI-CTCAE v4.0 grades. Laboratory abnormalities of NCI-CTCAE v4.0 Grades 3 and 4 are presented. Not every abnormal laboratory value qualified as an adverse event, only if it met any of the following criteria: clinically significant (per investigator); accompanied by clinical symptoms; resulted in a change in study treatment; or required a change in concomitant therapy. For the overall category, multiple occurrences of the same laboratory abnormality over time in one participant were only counted once.
Time Frame: Weeks 6, 12, and 18, and Unscheduled Visits (up to approximately 5 years)
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | Pertuzumab + Trastuzumab
Number analyzed (Participants) | 39
Participants
  Overall: Glucose (mmol/L), Low - Grade 3 | 0
  Overall: Glucose (mmol/L), High - Grade 3 | 2
  Overall: Glucose (mmol/L), Low - Grade 4 | 0
  Overall: Glucose (mmol/L), High - Grade 4 | 0
  Week 6: Glucose (mmol/L), High - Grade 3: number analyzed (Participants) | 30
  Week 6: Glucose (mmol/L), High - Grade 3 | 1
  Week 12: Glucose (mmol/L), High - Grade 3: number analyzed (Participants) | 26
  Week 12: Glucose (mmol/L), High - Grade 3 | 1
  Week 18: Glucose (mmol/L), High - Grade 3: number analyzed (Participants) | 22
  Week 18: Glucose (mmol/L), High - Grade 3 | 1
  Overall: Potassium (mmol/L), Low - Grade 3 | 0
  Overall: Potassium (mmol/L), High - Grade 3 | 0
  Overall: Potassium (mmol/L), Low - Grade 4 | 1
  Overall: Potassium (mmol/L), High - Grade 4 | 0
  Unscheduled Visit: Potassium (mmol/L),Low -Grade 4: number analyzed (Participants) | 10
  Unscheduled Visit: Potassium (mmol/L),Low -Grade 4 | 1

22. Secondary Outcome: Observed Trough Serum Concentrations (Cmin) of Pertuzumab at Specified Timepoints
Description: Per protocol eligibility criteria, participants were not required to be pertuzumab naïve; therefore pertuzumab was detectable in some participants pre-dose at Week 1.
Time Frame: Pre-dose (0-4 hours) on Day 1 of Weeks 1, 4, 10, and 16
Population: Pharmacokinetics (PK)-Evaluable Population: all participants who received any dose of study treatment and had at least one PK assessment unless there were major protocol deviations or if information impacting PK evaluation (e.g., exact blood sampling time, labeling error, technical failure in sample analysis) were unavailable.
Measure: Mean (Standard Deviation); unit: micrograms per millilitre (ug/mL)
Arm/Group | Pertuzumab + Trastuzumab
Number analyzed (Participants) | 39
micrograms per millilitre (ug/mL)
  Week 1 Day 1: number analyzed (Participants) | 38
  Week 1 Day 1 | 43.12 (101.45)
  Week 4 Day 1: number analyzed (Participants) | 33
  Week 4 Day 1 | 88.03 (29.91)
  Week 10 Day 1: number analyzed (Participants) | 32
  Week 10 Day 1 | 94.46 (38.47)
  Week 16 Day 1: number analyzed (Participants) | 22
  Week 16 Day 1 | 101.99 (41.59)

23. Secondary Outcome: Maximum Serum Concentrations (Cmax) of Pertuzumab at Specified Timepoints
Time Frame: Post-infusion (0-30 minutes, infused over 60 minutes) on Day 1 of Week 1 and 16
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: micrograms per millilitre (ug/mL)
Arm/Group | Pertuzumab + Trastuzumab
Number analyzed (Participants) | 39
micrograms per millilitre (ug/mL)
  Week 1 Day 1: number analyzed (Participants) | 35
  Week 1 Day 1 | 275.94 (88.80)
  Week 16 Day 1: number analyzed (Participants) | 22
  Week 16 Day 1 | 225.55 (56.22)

24. Secondary Outcome: Observed Trough Serum Concentrations (Cmin) of Trastuzumab at Specified Timepoints
Description: Per protocol eligibility criteria, participants were not required to be trastuzumab naïve; therefore trastuzumab was detectable in some participants pre-dose at Week 1.
Time Frame: Pre-dose (0-4 hours) on Day 1 of Weeks 1, 4, 10, and 16
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: micrograms per millilitre (ug/mL)
Arm/Group | Pertuzumab + Trastuzumab
Number analyzed (Participants) | 39
micrograms per millilitre (ug/mL)
  Week 1 Day 1: number analyzed (Participants) | 38
  Week 1 Day 1 | 57.00 (52.73)
  Week 4 Day 1: number analyzed (Participants) | 33
  Week 4 Day 1 | 190.82 (52.22)
  Week 10 Day 1: number analyzed (Participants) | 32
  Week 10 Day 1 | 294.50 (70.33)
  Week 16 Day 1: number analyzed (Participants) | 22
  Week 16 Day 1 | 306.14 (90.22)

25. Secondary Outcome: Maximum Serum Concentrations (Cmax) of Trastuzumab at Specified Timepoints
Time Frame: Post-infusion (0-30 minutes, infused over 60 minutes) on Day 1 of Week 1 and 16
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: micrograms per millilitre (ug/mL)
Arm/Group | Pertuzumab + Trastuzumab
Number analyzed (Participants) | 39
micrograms per millilitre (ug/mL)
  Week 1 Day 1: number analyzed (Participants) | 35
  Week 1 Day 1 | 181.43 (72.49)
  Week 16 Day 1: number analyzed (Participants) | 22
  Week 16 Day 1 | 394.14 (94.09)

26. Secondary Outcome: Symptom Severity Scale Score Over Time, Assessed by Participant Reporting on the M.D. Anderson Symptom Inventory-Brain Tumor (MDASI-BT) Questionnaire
Description: The MDASI-BT consists of 28 items and is a multi-symptom measure of cancer-related symptoms (Cleeland et al. 2000) that are sensitive to disease and treatment changes. The MDASI-BT is composed of the symptom severity scale and the symptom interference scale. In the symptom severity scale, participants rate the severity of their symptoms in the last 24 hours on 0-10 numeric scales, ranging from 0 = "not present" to 10 = "as bad as you can imagine." The MDASI-BT symptom severity scale score will be calculated by (sum of total scores of non-missing items) divided by (total number of non-missing items), if participants answered at least 12 of the 22 severity scale items. The score will be considered missing if less than 12 items are completed.
Time Frame: Baseline, Weeks 6, 12, 20, 28, 40, 52, and 64
Population: Patient-Reported Outcome (PRO)-Evaluable Population: all treated participants who had both a nonmissing baseline and at least one post-baseline PRO assessment.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Pertuzumab + Trastuzumab
Number analyzed (Participants) | 36
Score on a scale
  Baseline | 1.65 (1.618)
  Week 6: number analyzed (Participants) | 27
  Week 6 | 1.97 (1.822)
  Week 12: number analyzed (Participants) | 26
  Week 12 | 2.24 (2.141)
  Week 20: number analyzed (Participants) | 15
  Week 20 | 2.09 (2.111)
  Week 28: number analyzed (Participants) | 11
  Week 28 | 1.94 (2.547)
  Week 40: number analyzed (Participants) | 7
  Week 40 | 2.78 (2.856)
  Week 52: number analyzed (Participants) | 5
  Week 52 | 3.53 (3.018)
  Week 64: number analyzed (Participants) | 5
  Week 64 | 3.12 (2.500)

27. Secondary Outcome: Symptom Interference Scale Score Over Time, Assessed by Participant Reporting on the MDASI-BT Questionnaire
Description: The MDASI-BT consists of 28 items and is a multi-symptom measure of cancer-related symptoms that are sensitive to disease and treatment changes. The MDASI-BT is composed of the symptom severity scale and the symptom interference scale. In the symptom interference scale, participants rate interference with daily activities caused by their symptoms on 0-10 numeric scales ranging from 0 = "did not interfere" to 10 = "interfered completely." The MDASI-BT symptom interference scale score will be calculated by (sum of total scores of non-missing items) divided by (total number of non-missing items), if participants answered at least 4 of the 6 interference scale items. The score will be considered missing if less than 4 items are completed.
Time Frame: Baseline, Weeks 6, 12, 20, 28, 40, 52, and 64
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Pertuzumab + Trastuzumab
Number analyzed (Participants) | 36
Score on a scale
  Baseline | 2.51 (2.629)
  Week 6: number analyzed (Participants) | 27
  Week 6 | 2.23 (2.787)
  Week 12: number analyzed (Participants) | 24
  Week 12 | 2.81 (3.391)
  Week 20: number analyzed (Participants) | 15
  Week 20 | 2.11 (2.858)
  Week 28: number analyzed (Participants) | 11
  Week 28 | 1.76 (2.427)
  Week 40: number analyzed (Participants) | 7
  Week 40 | 3.24 (3.548)
  Week 52: number analyzed (Participants) | 5
  Week 52 | 4.25 (3.522)
  Week 64: number analyzed (Participants) | 5
  Week 64 | 3.93 (3.570)

ADVERSE EVENTS:
Time Frame: From first dose of study drug until 30 days after last dose of study drug (except for serious AEs related to treatment; up to approximately 5 years)
Description: Investigators seek information on adverse events (AEs) at each patient contact. All AEs were recorded, regardless of who reported them. After informed consent but prior to initiation of study drug, only serious AEs caused by protocol-mandated intervention were to be reported. After initiation of study drug, all AEs were to be reported until 30 days after the last dose of study drug. After this period, only serious AEs believed to be related to prior study drug treatment were to be reported.
Arm/Group | Pertuzumab + Trastuzumab
All-Cause Mortality (participants affected / at risk) | 20/39
Serious Adverse Events (participants affected / at risk) | 7/39
Other Adverse Events (participants affected / at risk) | 38/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pertuzumab + Trastuzumab (N=39)
Gastroenteritis viral (Infections and infestations) | 1 (1)
Parainfluenzae virus infection (Infections and infestations) | 1 (1)
Seizure (Nervous system disorders) | 4 (4)
Headache (Nervous system disorders) | 1 (1)
Hydrocephalus (Nervous system disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pertuzumab + Trastuzumab (N=39)
Anaemia (Blood and lymphatic system disorders) | 3 (3)
Vision blurred (Eye disorders) | 4 (6)
Diarrhoea (Gastrointestinal disorders) | 23 (30)
Nausea (Gastrointestinal disorders) | 12 (21)
Vomiting (Gastrointestinal disorders) | 12 (16)
Constipation (Gastrointestinal disorders) | 7 (9)
Dry mouth (Gastrointestinal disorders) | 3 (4)
Dysphagia (Gastrointestinal disorders) | 4 (4)
Abdominal distension (Gastrointestinal disorders) | 2 (6)
Abdominal pain (Gastrointestinal disorders) | 2 (5)
Dyspepsia (Gastrointestinal disorders) | 3 (5)
Stomatitis (Gastrointestinal disorders) | 2 (2)
Fatigue (General disorders) | 17 (21)
Asthenia (General disorders) | 6 (6)
Gait disturbance (General disorders) | 5 (5)
Pain (General disorders) | 4 (4)
Mucosal inflammation (General disorders) | 3 (3)
Oedema peripheral (General disorders) | 2 (5)
Upper respiratory tract infection (Infections and infestations) | 6 (10)
Urinary tract infection (Infections and infestations) | 5 (11)
Gastroenteritis viral (Infections and infestations) | 2 (2)
Nasopharyngitis (Infections and infestations) | 2 (2)
Sinusitis (Infections and infestations) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 4 (7)
Contusion (Injury, poisoning and procedural complications) | 3 (3)
Infusion related reaction (Injury, poisoning and procedural complications) | 3 (3)
Alanine aminotransferase increased (Investigations) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 3 (3)
Blood alkaline phosphatase increased (Investigations) | 2 (2)
Neutrophil count decreased (Investigations) | 2 (5)
Platelet count decreased (Investigations) | 2 (2)
Weight increased (Investigations) | 2 (3)
White blood cell count decreased (Investigations) | 2 (4)
Decreased appetite (Metabolism and nutrition disorders) | 6 (6)
Hypokalaemia (Metabolism and nutrition disorders) | 6 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (8)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 (5)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (5)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Dizziness (Nervous system disorders) | 7 (10)
Headache (Nervous system disorders) | 6 (15)
Paraesthesia (Nervous system disorders) | 4 (7)
Dysarthria (Nervous system disorders) | 3 (3)
Neuropathy peripheral (Nervous system disorders) | 3 (3)
Syncope (Nervous system disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 7 (7)
Anxiety (Psychiatric disorders) | 5 (5)
Depression (Psychiatric disorders) | 2 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (5)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (5)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Rash (Skin and subcutaneous tissue disorders) | 6 (7)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (7)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2)
Rash papular (Skin and subcutaneous tissue disorders) | 2 (2)
Hypertension (Vascular disorders) | 3 (4)
Hot flush (Vascular disorders) | 2 (2)
Ear pain (Ear and labyrinth disorders) | 2 (2)
Dry eye (Eye disorders) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2)
Rectal haemorrhage (Gastrointestinal disorders) | 2 (2)
Pyrexia (General disorders) | 2 (2)
Swelling face (General disorders) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Memory impairment (Nervous system disorders) | 2 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2)
Taste disorder (Nervous system disorders) | 2 (4)
Seizure (Nervous system disorders) | 2 (2)
Vaginal haemorrhage (Reproductive system and breast disorders) | 2 (2)
Onychoclasis (Skin and subcutaneous tissue disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2018-10-29): https://cdn.clinicaltrials.gov/large-docs/39/NCT02536339/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-29): https://cdn.clinicaltrials.gov/large-docs/39/NCT02536339/SAP_001.pdf